CLINICAL TRIAL: NCT05811676
Title: Department of Obstetrics and Gynecology, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, PR China
Brief Title: Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Pregnant Women With Placenta Previa
Acronym: TRAPP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Collaborators: Dongguan Maternal and Child Health Care Hospital (Unknown); Foshan Women's and Children's Hospital (Other); BoAi Hospital of Zhongshan (Other); Women and Children's Hospital of Chongqing Medical University (Unknown); Tianjin Central Hospital of Gynecology Obstetrics (Other); Shandong Provincial Maternal and Child Health Care Hospital Affiliated to Qingdao University, Jinan (Unknown); Urumqi Maternal and Child Health Care Hospital (Unknown); Zhuhai Women and Children's Hospital (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); Dalian women and children's medical group (Unknown); Nanfang Hospital, Southern Medical University (Other); Huadu District People's Hospital of Guangzhou (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Shenzhen Maternity & Child Healthcare Hospital (Other); Shenzhen Baoan Women's and Children's Hospital (Unknown); Dongguan People's Hospital (Other Government); First Affiliated Hospital of Xinjiang Medical University (Other); Tongji Hospital (Other); Peking Union Medical College (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Shijiazhuang Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Dunjin Chen, Department of Obstetrics and Gynecology, The Third Affiliated Hospital, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MR-44-23-016012（TRAPP）
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-08

CONDITIONS: Hemorrhage, Postpartum; Placenta Previa
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Previa | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): Intravenous administration of 10 mL (1 g of tranexamic acid) diluted in 40 ml of normal saline, over 10 minutes after umbilical-cord clamping, the routine prophylactic uterotonic administration
  Interventions: Drug: Tranexamic acid
- control group (Placebo Comparator): Intravenous administration of 10 mL placebo (0.9% sodium chloride), diluted in 40 ml of normal saline, over 10 minutes after umbilical-cord clamping, the routine prophylactic uterotonic administration
  Interventions: Other: 0.9% sodium chloride

INTERVENTIONS:
Drug: Tranexamic acid — Intravenous administration of 10 mL (1 g of tranexamic acid), diluted in 40 ml of normal saline, over 10 minutes after umbilical-cord clamping, the routine prophylactic uterotonic administration
  Arms: study group
Other: 0.9% sodium chloride — Intravenous administration of 10 mL placebo(0.9% sodium chloride), diluted in 40 ml of normal saline, over 10 minutes after umbilical-cord clamping, the routine prophylactic uterotonic administration
  Arms: control group

SUMMARY:
Many RCT(randomized controlled trial) studies reported that tranexamic acid reduced blood loss in women who had elective cesareans. However, most of these elective cesareans are without high-risk factors of postpartum hemorrhage, such as placenta previa. The prophylactic use of tranexamic acid in the placenta previa is not clear.

studies had poor quality and lacked adequate power to assess severe adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Diagnosed with Placenta previa before cesarean delivery by ultrasound（Placenta previa defined by a placental edge below 20mm from internal cervical os diagnosed at the most recent transvaginal ultrasound examination before delivery）
* Gestational age ≥ 34 weeks
* Available venous hematocrit value in the week before the cesarean
* Prenatal hemoglobin level in the week before the cesarean > 90 g/l
* Undergoing cesarean delivery
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to tranexamic acid or concentrated hydrochloric acid
* History of venous (deep vein thrombosis and/or pulmonary embolism) or arterial thrombosis (angina pectoris, myocardial infarction, or stroke)
* History of epilepsy or seizure
* Any known active cancer, active cardiovascular, renal, or liver disorders
* Autoimmune diseases such as lupus, rheumatoid arthritis, Sjogren's disease, and inflammatory bowel disease
* Sickle cell disease
* Severe hemorrhagic disease
* Administration of low-molecular-weight heparin or antiplatelet agents within one week prior to delivery
* Severe coagulation disorders with prothrombin time or activated partial thromboplastin time exceeding the upper limit of normal, or platelet count less than 80×109/L
* placenta abruption
* In-utero fetal death
* Eclampsia or HELLP syndrome
* Acquired color vision deficiency or subarachnoid hemorrhage
* Severe bleeding with estimated blood loss exceeding 500 ml, within 12 hours before cesarean delivery
* Known congenital or acquired thrombophilias, including antiphospholipid antibody syndrome
* Participation in another intervention study where the primary outcome includes postpartum bleeding or thromboembolism or the study intervention potentially affects postpartum bleeding or thromboembolism

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1732 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-03-23 (Actual)

PRIMARY OUTCOMES:
Incidence of PPH | Day 2
  defined by a calculated estimated blood loss > 1000 mL [Calculated estimated blood loss = estimated blood volume × (preoperative hematocrit - postoperative hematocrit)/preoperative hematocrit (where estimated blood volume (mL) = weight (Kg) × 85)] or red blood cell (RBC) transfusion before day 2 postpartum .

SECONDARY OUTCOMES:
mean total calculated blood loss | Day 2
  Calculated estimated blood loss = estimated blood volume × (preoperative hematocrit - postoperative hematocrit)/preoperative hematocrit (where estimated blood volume (mL) = weight (Kg) × 85)] or red blood cell (RBC) transfusion before day 2 postpartum
mean gravimetrically estimated blood loss | postpartum 24 hours
  estimated blood loss = (weight of materials used + materials not used - weight of all materials before surgery)/ 1.05 + volume included in the suction container
Number of Participants with additional uterotonic agents treatment | baseline
  additional uterotonic agents include oxytocin, carbetocin, carboprost, misoprostol, ergonovine et al
incidence of postpartum transfusion | baseline
  include RBC, plasma, platelet, cryo et al
incidence of postpartum iron perfusion | baseline
incidence of hypovolemic shock related to PPH | baseline
incidence of interventional therapy | baseline
  include arterial embolization, abdominal aortic balloon, internal iliac artery/common iliac artery balloon et al
incidence of transfer to intensive care unit | baseline
Number of Participants with additional operations performed outside cesarean section | baseline
  Additional operations include B-Lnych, uterine artery suture, partial hysterectomy, hysterectomy et al
incidence of maternal death from any cause | week 6
incidence of hospital readmission | baseline
mean peripartum change in hemoglobin | Day 2
  the difference between the hemoglobin levels before delivery and at D2
mean peripartum change in hematocrit levels | Day 2
  the difference between the hematocrit levels before delivery and at D2
incidence of infectious complications | week 6
  include endometritis, surgical-site infection, or pelvic abscess within 6 weeks post partum
incidence of maternal thromboembolic events | week 6
  including venous, arterial, or ischemic stroke or myocardial infarction within 6 weeks post partum

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - Department of Obstetrics and Gynecology, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking Union Medical College, Beijing
  - Peking University First Hospital, Beijing
  - Women and Children's Hospital of Chongqing Medical University, Chongqing
  - Dalian Women and Children's Medical Group, Dalian
  - Dongguan Maternal and Child Health Care Hospital, Dongguan
  - The Tenth Affiliated Hospital of Southern Medical University; Dongguan People's Hospital, Dongguan
  - Foshan Women and Children Hospital, Foshan
  - Boai Hospital of Zhongshan, Guangzhou
  - Huadu District People's Hospital of Guangzhou, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangzhou
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The first Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhuhai Women and Children's Hospital, Guangzhou
  - Obstetrics Department, the Maternal and Child Health Hospital of Hunan Province, Hunan
  - Shandong Provincial Maternal and Child Health Care Hospital Affiliated to Qingdao University, Jinan
  - Shenzhen Baoan Women's and Children's Hospital, Shenzhen
  - Shenzhen Maternal ＆ Child Healthcare Hospital Affiliated Southern Medical University, Shenzhen
  - Shijiazhuang Obstetrics and Gynecology Hospital, Shijiazhuang
  - Tianjin Central Hospital of Gynecology Obsterics, Tianjin
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Northwest Women's and Children's Hospital, Xi'an
  - First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Urumqi Maternal and Child Health Care Hospital, Xinjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

REFERENCES:
- [Derived] Zhang L, Hu M, Bi S, Poon LC, He F, Li H, Zhang Y, Gu Z, Wang Z, Du L, Chen D; TRAPP Study Group. TRAPP- Protocol for Tranexamic Acid for the Prevention of Postpartum Hemorrhage in Pregnant Women With Placenta Previa. Matern Fetal Med. 2026 Jan;8(1):3-12. doi: 10.1097/FM9.0000000000000297. Epub 2025 Jul 15. PMID 41624591